CLINICAL TRIAL: NCT05265143
Title: Comparision of Two Different Feeding Method in Preterm Infants
Brief Title: Comparision of Two Different Feeding Method in Preterms
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zekai Tahir Burak Women's Health Research and Education Hospital (Other)
Responsible Party: Principal Investigator, Funda Yavanoglu Atay, principal investigator, Zekai Tahir Burak Women's Health Research and Education Hospital
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Other
Other Study IDs: 2579
Record Dates: First submitted 2022-02-09; First posted 2022-03-03 (Actual); Last update posted 2022-03-03 (Actual); Status verified 2022-02

CONDITIONS: Enteral Feeding Intolerance
Keywords: preterm; feeding intolerence
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- bolus feeding group (Other): In bolus feednig group preterm fed by via gravity drip over a short period, usually 15-20 min. it administrated 8-12 times daily
  Interventions: Other: bolus/intermittant feeding
- intermittant feeding group (Other): Intermittant feeding is delivered over a 30-60 min by infusion pump. it administrated 8-12 times daily
  Interventions: Other: bolus/intermittant feeding

INTERVENTIONS:
Other: bolus/intermittant feeding — sequential randomization

SUMMARY:
achievement of optimal postnatal growth by adequate enteral nutrition in critically ill preterm infants is a challenge of NICU. signs like abdominal distension, reflux, vomiting, nec is a factors of discontinuing fedding in preterm. this factors plays a role in decisions about which method of gavage feeding is adopted. we compare two different feeding method to achive less fedding tolerence.

DETAILED DESCRIPTION:
<1750 gr, <33 gw infants will enroll study. exckusion criteria: major congenital anomalies major gis anomalies

The study infants are enrolled within 24 hours of birth and sequently randomized to either intermitten feeding (IF) and bolus feeding (BF). Intermittent feeding is defined as delivering enteral nutrition and generally giving 60 min and 2 hours no feeding. this circle repeats 8 times in 24 hours. Bolus feeding is the amount of nutrition put into the syringe was kept 10 cm above the baby and the fluidity was obtained by gravity through the orogastric tube. The data of the patients such as feeding intolerance (gastric residual volume more than %50 of the previous feeding volume, gastric regurgitation, abdominal distension and/or emesis ), whether there is a week-by-week feeding intolerance were noted, NEC, time to reached birth weight, time to achieved full enteral feeding, every 5 minutes during feeding, saturation, respiratory rate and heart rates will record.

ELIGIBILITY:
Inclusion Criteria:

* <1750 gr preterm infants
* <33 gw
* admitted to our nicu in first day of life

Exclusion Criteria:

major congenital anomalies gis anomalies septic shock exitus in 3 days of life

-

Ages: 1 Day to 3 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 100 (Estimated)
Dates: Start 2015-01-01 (Actual); Primary Completion 2022-06-01 (Estimated); Study Completion 2022-06-01 (Estimated)

PRIMARY OUTCOMES:
rate of feeding intolerence | 1 month
  The effect of two different gavage tube feeding methods on feeding intolerance

SECONDARY OUTCOMES:
time to reach full enteral feeding | 1 month
  The effect of two different gavage tube feeding methods on time to reach full enteral feeding

CONTACTS AND LOCATIONS:
Overall Officials: Funda Yavanoğlu Atay, md, Principal Investigator — Zekai Tahir Burak Women's Health Research and Education Hospital
Locations (1):
- Ümraniye Teaching Hospital, Istanbul, Turkey (Türkiye)

REFERENCES:
- [Background] Richards R, Foster JP, Psaila K. Continuous versus bolus intermittent intragastric tube feeding for preterm and low birth weight infants with gastro-oesophageal reflux disease. Cochrane Database Syst Rev. 2021 Aug 6;8(8):CD009719. doi: 10.1002/14651858.CD009719.pub3. PMID 34355390